CLINICAL TRIAL: NCT01344330
Title: Cruciferous Vegetable Intake and Histone Status in Screening Colonoscopy Patients
Status: Completed | Type: Observational
Sponsor: Texas A&M University (Other)
Collaborators: Oregon Health and Science University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roderick Dashwood, Professor, Texas A&M HSC, Texas A&M University
Other Study IDs: P01CA090890 (NIH); P01CA090890 (NIH)
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Prevention; Cruciferous vegetables; Histone status
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Protein lysate and RNA obtained from de-identified normal colon biopsy specimens are stored at -80 degree centigrade.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Screening colonoscopy patients: Men and women age 50 to 75 scheduled for screening colonoscopy

SUMMARY:
This research study will assess cruciferous vegetable intake in patients presenting for screening colonoscopy and correlate intake with histone status and histone deacetylace (HDAC) expression in tissue biopsy specimens and peripheral blood mononuclear cells (PBMCs). The investigators will also measure sulforaphane (SFN) metabolites in blood as a biomarker of cruciferous vegetable intake.

ELIGIBILITY:
Inclusion criteria:

* scheduled for screening colonoscopy
* off NSAID or aspirin therapy in accordance with OHSU endoscopy clinic guidelines
* INR 0.90-1.20
* hemoglobin ≥ 13.5 (men) or 12.0 (women)
* platelets ≥100,000/μL
* Chem screen results within normal limits
* negative (serum or urine) pregnancy test done ≤7 days prior to colonoscopy for women of childbearing potential only
* ASA performance status <2

Exclusion criteria:

* history of colon cancer or adenomatous polyps
* current smoker
* medical history of chronic obstructive pulmonary disease
* current oral steroid therapy
* current therapy with valproate or other pharmacological drugs associated with HDAC inhibition
* use of oral antibiotics within 3 months prior to entry into study
* significant active medical illness which in the opinion of the investigator would preclude collection/interpretation of colon tissue
* diagnosis of hemophilia, van Willebrand's disease or other bleeding disorder
* use of warfarin or other blood thinning agents
* inflammatory bowel disease.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for screening colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cruciferous vegetable intake correlated with SFN and I3C urinary metabolites | At colonoscopy (day 1)

SECONDARY OUTCOMES:
Cruciferous vegetable intake and p21 expression (qRT-PCR, ChIP in PBMCs) | at colonoscopy
Cruciferous vegetable intake correlated with acetylated histone expression (PBMCs, colon tissue), | at colonoscopy
Cruciferous vegetable intake correlated with HDAC activity (in PBMCs) | at colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Rod Dashwood, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Group information (High versus Low Cruciferous Vegetable Intake) will be made available. No IPD will be made available.